# TITLE: CLINICAL PHARMACOLOGY OF ELECTRONIC CIGARETTES

## NCT02470754

Date: 4/15/2019

#### **Abbreviations**

**EC** Electronic Cigarette

TC Tobacco Cigarette (Commercially Manufactured or Available)

PK Pharmacokinetic
CI Confidence Interval
SD Standard Deviation

BMI Body Mass Index

HR Heart Rate

SBP Systolic Blood Pressure
DBP Diastolic Blood Pressure

**hr** Hour

**AUCinf** Area under the plasma concentration time curve from zero to the last measured time

AUClast Area under the plasma concentration time curve extrapolated from zero

CMAX Peak Plasma Concentration

**TMAX** Time of Peak Plasma Concentration

**THalf** Half-Life

ANOVA Analysis of Variance SAS Statistical Analysis System

## **Study Design**

This is a within-subject two-arm crossover study design evaluating the safety and addictive potential of EC compared to TC



| Study Block #2 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Day #1 | Day #2 | Day #3 | Day #4 | Day #5 | Day #6 | Day #7 | Day #8 | Day #9 |
| ı | Thursday | Friday | Saturday | Sunday | Monday | Tuesday | Wednesday | Thursday | Friday |
| ı | Outpatient | Outpatient | Outpatient | Outpatient | Inpatient | Inpatient | Inpatient | Inpatient | Inpatient |
| l | | | | | | | | | |
| ı | Blood Draw | | | | | Ad lib use | Ad lib use | Abstinence | Abstinence |
| ı | Urine Collection | | | | Single Use PK | 24-hr CV monitoring | Circadian Bloods | 24-hr CV monitoring | 24-hr CV monitoring |
| ı | Aller Control of the | D/Cin AM Ad lib use of | | | | 24-hr Urines | 24-hr Urines | 24-hr Urines | 24-hr Urines |
| w/ 2nd study<br>product | | dispensed | | | Questionnaires | Questionnaires | Questionnaires | Questionnaires | Questionnaires |
| ١ | + | study product | | - | | | | | Blood Draw |
| ı | | | | | | | | | |

#### **Study Endpoints**

On the first hospital day in each treatment arm the subject will use their product at 9 AM in a standardized protocol. EC use will be one puff every puff every 30 seconds for a total of 15 puffs on 1st generation devices and 10 puffs on 2nd/3rd generation devices.

Endpoint (s): Systemic Nicotine Exposure - Baseline Adjusted AUC (Inf), TMAX, CMAX, Half-Life, and PK-Predicted Dose following the standardized puffing protocol. Additional PK Parameters may be calculated as deemed necessary.

Analysis: Linear mixed model

Descriptive Summary Statistics: N, n, arithmetic mean, SD, 95% CI will be used to describe continuous measures including nicotine intake [AUC Inf, AUC Last, PK-predicted dose] related to single use PK. Categorical Data will be described using frequency count and percentage of subjects in each category. Descriptive statistics will be calculated using standard methods.

#### **Statistical Hypothesis**

Distributional assumptions underlying the model will be examined by analysis of the residuals and plot of the residuals vs the fitted values.

Treatment effects will be compared by means of repeated measures ANOVA. All significance tests will be two-sided with an alpha level set at 0.05.

#### **Primary Analysis**

Crossover analysis was carried out following standard procedures. Following In-transformation of plasma concentrations treatment effects were compared by means of repeated measures ANOVA. To account for the relatedness in the plasma nicotine measures within each subject during the two treatment periods, a linear mixed model was used to account for non-independence in sequential measurements. In building the linear mixed-models, baseline-adjusted plasma nicotine concentrations were considered the dependent variable. These models included independent variables of treatment and a dichotomized variable defining order of product assignment. Participant IDs were used as group factor to estimate random effects.

## **Secondary Analysis**

PK data will be presented in graphical and/or tabular form and will be summarized descriptively. Mean Heart Rate, Mean Systolic Blood Pressure and Mean Diastolic Blood Pressure will also be described similarly. Additional toxicant exposure data may be described as necessary.